CLINICAL TRIAL: NCT05545241
Title: Awareness of Emotional Feelings and Management of Risky Situations
Acronym: COSMOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Plateforme Neuraxess (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022/718
Record Dates: First submitted 2022-09-08; First posted 2022-09-19 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Risk-Taking; Emotional Regulation
Keywords: risk-taking; emotional neurofeedback; emotional regulation
MeSH Terms: conditions — Risk-Taking; Emotional Regulation | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurofeedback and BART-EEG assessment (Experimental): Healthy subjects realized 10 sessions of emotional neurofeedback. Before (Baseline, Day 0), and after (at the study completion (after 10 neurofeedback sessions, Week 5)) neurofeedback sessions, the BART, assessing risk-taking behavior, coupled with an EEG record is realized by the subjects.
  Interventions: Behavioral: Neurofeedback + BART/EEG
- BART-EEG assessment without neurofeedback (Sham Comparator): At the same times (Baseline, Day 0), and at the study completion (after 10 neurofeedback sessions, Week 5), healthy subjects realized the BART, assessing risk-taking behavior, coupled with an EEG record.
  Interventions: Behavioral: BART/EEG only

INTERVENTIONS:
Behavioral: Neurofeedback + BART/EEG — 10 sessions of emotional neurofeedback (max of 2 sessions per week and max of 10 weeks).
  Before (Baseline, Day 0) and at the study completion (after 10 neurofeedback sessions, Week 5), a EEG record is realized during the BART, assessing risk-taking behavior.
  Arms: Neurofeedback and BART-EEG assessment
Behavioral: BART/EEG only — only the twice EEG record are realized during the BART, assessing risk-taking behavior (every corresponding to the pre and post-neurofeedback evaluations in arm I)
  Arms: BART-EEG assessment without neurofeedback

SUMMARY:
The goal of this project is to help individuals better self-assess by taking advantage of their emotional feelings.

DETAILED DESCRIPTION:
All emotions such as sadness, anger, fear or joy undoubtedly have an important place in our lives. Our emotions influence all areas of our lives and particularly our relationships: with our spouses, our friends, our children, our colleagues. Emotions are necessary for our decisions. By influencing our decisions, emotions automatically impact our performance.

By guiding our choices, our emotions lead us to take risks. Taking risks is sometimes essential to a suitable decision. But this risk-taking must not result from an inappropriate decision-making process. People must therefore adapt their risk-taking, i.e. integrate our emotions into decision-making. It is therefore not a question of ignoring one's emotions, but of regulating them in order to be in a state favorable to action. This awareness of emotional feelings would help develop the ability to produce good internal feedback.

The purpose of COSMOS project is to help individuals better self-assess by taking advantage of their emotional feelings. To do this, investigators will teach individuals to detect and manage their emotions using an emotional neurofeedback device developped by the Neuraxess platform (a functional neuroimiaging and neurostimulation platform, located in Besancon, France). Neurofeedback is a type of biofeedback, namely a rehabilitation method based on the subject's awareness of physiological processes, during which the neuronal activity of an individual is measured and presented to him in real time, here in artistic form. The goal of this method is that the individual manages to self-regulate his neuronal activity supposed to underlie a specific behavior. So, over time, the participant might be able to learn how to voluntarily control the activation of their cerebral cortex in order to regulate their emotions and behaviors in everyday life. Here, by learning to detect and manage their emotions, participants will be able to take more appropriate risks. The balloon test (Balloon Analogue Risk Task or BART) is used to measure risk taking. This tasks consists of inflating a balloon by clicking on a button on the computer. The more the balloon inflates, the more money participants earn, but the involved risk is to reach a threshold where the balloon bursts and participants lose everything. Participants have the choice between reaching the limit and losing everything or controlling ourselves and recovering our gains before the disaster. This is a simple test but it closely matches the behavior of the player at a poker or roulette table in a casino. Participants' risk-taking will be assessed before the emotional neurofeedback sessions and then after 10 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 80 years old
* Right-handed
* Signed informed Consent Form
* Subject affiliated to or beneficing from a French social security regime

Exclusion Criteria:

* Subjects under 18 years old and over 80 years old
* Left-handed
* Pregnant woman
* Subject beneficiary from a legal protection regime
* Subject unlikely to cooperate or low cooperation stated by investigator
* Subject not covered by social security
* Subject being in the exclusion period of another study or provided for by the "National Volunteer File"

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in number of blue balloons adjusted with Balloon Analogue Risk Task [BART] | Baseline (Day 0), at the study completion (after 10 neurofeedback sessions, Week 5)
  Number of blue balloons adjusted with BART after 10 neurofeedback sessions among participants who received the neurofeedback treatment.

SECONDARY OUTCOMES:
Change in EPs during BART | Baseline (Day 0), at the study completion (after 10 neurofeedback sessions, Week 5)
  Amplitude variation of evoked potentials (EPs) detected by electroencephalography (EEG) during the Balloon Analogue Risk Task (BART), assessing risk-taking behavior. Variation will be obtained by comparing records before and after 10 neurofeedback sessions
Feasibility of controlling brain activity during neurofeedback sessions | Baseline (Day 0), immediately after each neurofeedback sessions (session 1 to session 10) and at the study completion (after 10 neurofeedback sessions, Week 5)
  Satisfaction assessed by a visual analogue scale (items: "I enjoyed participating in the experiment" ; "I was motivated during the experience" ; "I managed to control the particles by thought" and "I feel more relaxed after session".
Change in BIS-10 scores | Baseline (Day 0), at the study completion (after 10 neurofeedback sessions, Week 5)
  Compared scores from the French version of the Barratt Impulsiveness Scale (BIS-10). The French version of the BIS-10 is a self-rated 34 item questionnaire, composed by three subscales: motor-impulsivity, cognitive-impulsivity and non-planning-impulsivity. Each item is scored on a 0 to 4 points scale. Higher scores indicate higher levels of impulsivity.
Change in MCQ scores | Baseline (Day 0), at the study completion (after 10 neurofeedback sessions, Week 5)
  Compared scores from the French version of the Monetary Choice Questionnaire (MCQ). The MCQ is a self-rated 27 item questionnaire which assessed the discounting. Delay discounting is the decline in the present value of a reward with delay to its receipt.
  Example item: " Would you prefer 25€ today or 75€ in 15 days? " For each item, subjects must choose between a low immediate reward and a higher delayed reward.
  Waiting times vary from 7 days to 186 days, and rewards are divided into 3 magnitudes: low (25-35€), medium (50-60€), high (75-85€).
  This will allow assessing: the influence of the the magnitude of the difference between the two rewards proposed, the impact of the time on the reward's subjective value (speed at which the reward is devalued over time), reflected in the k index.
  This index is calculated separately for each magnitude, and an average index is calculated for each subject.
  The more the k index is high, the more the subject is considered impulsive.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besancon - Clinical Psychiatric Department, Besançon, France